CLINICAL TRIAL: NCT06373536
Title: Comparison of Thermoacoustic Enhanced Ultrasound for Estimating Liver Fat Fraction to MRI-PDFF
Brief Title: Comparison of MRI-PDFF to TAEUS FLIP Device to Estimate Liver Fat Fraction in Adults
Status: Not yet recruiting | Type: Observational
Sponsor: Endra Lifesciences (Industry)
Responsible Party: Sponsor
Other Study IDs: LMU-RAD-01167
Record Dates: First submitted 2024-04-05; First posted 2024-04-18 (Actual); Last update posted 2024-06-07 (Actual); Status verified 2024-04

CONDITIONS: Steatosis of Liver
Keywords: MRI-PDFF; Thermoacoustics
MeSH Terms: conditions — Fatty Liver | interventions — Magnetic Resonance Imaging; Ultrasonography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Thermoacoustic imaging, MRI and Ultrasound imaging — This is a Thermoacoustic imaging exam that will last 10-15 minutes. Distinguishing; assessment of steatosis liver disease in obese and morbidly obese patients.

SUMMARY:
Primary nonalcoholic fatty Liver disease (NAFLD) is an excess of fat in the liver (steatosis) that is not a result of excessive alcohol consumption or other secondary causes11. NAFLD is defined by the presence of hepatic fat content (steatosis) in ≥ 5% of hepatocytes and is currently the most common liver disease worldwide14 . Non-Alcoholic Fatty Liver Disease (NAFLD) is the world's most common liver disease and affects around 33% of the adult population.

Nonalcoholic steatohepatitis (NASH), a progressive form of nonalcoholic fatty liver disease (NAFLD), is a growing clinical concern associated with the increasing prevalence of obesity, type 2 diabetes, and metabolic syndrome. NASH is characterized by the presence of hepatic steatosis, inflammation, and hepatocellular injury and is predicted to be the leading indication for liver transplantation by 20201. Patients with NASH have an increased risk of developing cirrhosis and its complications, such as ascites, variceal hemorrhage, hepatic encephalopathy, hepatocellular carcinoma, and liver failure. The prevalence worldwide of NAFLD in the general population is estimated at 20-35%2 . Around 2-3% of the population have NASH.

In patients with type 2 diabetes, the prevalence is even over 50% (55.5% globally, 68% in Europe). In Germany, the NAFLD prevalence was 23% in 2016 and will be around 26% in 2030. The prevalence of non-alcoholic alcoholic steatohepatitis (NASH), i.e. the progressive form of NAFLD, is estimated at 4% of the adult population in Germany and will increase to 6% by 2030. This means that NAFLD is already the most common chronic liver disease worldwide and one of the leading causes of liver-related complications (cirrhosis, decompensation, hepatocellular carcinoma, liver transplantation) and deaths. NAFLD and NASH are largely underdiagnosed worldwide.

DETAILED DESCRIPTION:
Early detection and surveillance of steatosis hepatis improves the chances of management or even improvement of the disease before irreversible damage occurs12. Liver tissue biopsy is the current reference standard for the diagnosis and severity of steatosis hepatis. However, due to its invasiveness, biopsy collection is not suitable for screening or regular follow-up. The diagnostic techniques of magnetic resonance spectroscopy (MRS) and MRI-PDFF (proton density fat fraction) for the assessment of liver fat content have been shown to correlate well with the results of liver biopsy, but are particularly associated with high costs, low availability, long examination times and exclusion of patients with metal implants. Conventional B-scan ultrasonography is the most commonly used imaging modality for assessing steatosis hepatis based on qualitative image features of the liver. These include an echo-enhanced internal reflex pattern of the liver parenchyma, loss of signal in depth, blurred demarcation of the blood vessels and diaphragm, or areas of focal obesity. The sensitivity and specificity of conventional sonography is high in severe steatosis hepatis. On the other hand, the sensitivity is significantly worse in mild cases. In addition, intra- and interobserver reliability are poor in the assessment of steatosis hepatis of the conventional B-scan.

Quantitative ultrasound-based methods are the current standard of practice for point-of-care, noninvasive liver fat assessment. However, due to low penetration depth and confounding factors, invalid or poor-quality measurements are often encountered in large patients, or patients with liver fibrosis. In contrast to purely ultrasound-based approaches, thermoacoustic (TA) approaches are sensitive to tissue composition chemistry rather than acoustic scattering and/or attenuation, making TA measurements of liver fat content relatively insensitive to liver fibrosis or patient size.

Thermoacoustic (imaging) technology is non-invasive and combines short pulses of radio-frequency energy to create ultrasound signals (acoustic waves) in tissue to create images, or measurements, of fat in body tissues. The radio-frequency energy that is used to create thermoacoustic ultrasound signals is very similar to that used by cell phones and MRI scanners. Thermoacoustic signals are created in proportion to how well tissue is able to conduct electricity. Lean tissues are highly conductive while fatty tissues are not, and thus, thermoacoustics is able to differentiate lean and fatty tissues. A primary interest in detecting, and monitoring metabolic health, is measuring liver fat content. Thermoacoustic approaches to fat measurement in the liver have several unique advantages compared to other currently used technologies, including ultrasound and MRI. Medical ultrasound scanners are widely available but often have difficulty making high-quality images, and reliable measurements, in larger patients or deeper tissues. Thermoacoustic ultrasound signals are formed in the tissue allowing measurements of fat to be made at depths that may not be possible with conventional ultrasound systems. While MRI is the most accurate noninvasive method to estimate fat in tissue, it has limited availability and is very expensive compared to thermoacoustics, and thus impractical for widespread use that is needed to address the growing problem of fatty liver disease and metabolic syndrome.

Thermoacoustic approaches to fat measurement in tissue are exceptionally safe using radio frequency energy levels similar to MRI, with tissue heating that is less than a 0.001 degrees Celsius per pulse in temperature. ENDRA has developed a noninvasive bedside device called the TAEUS®-FLIP system for measuring fat in liver tissue. The TAEUS®-FLIP exam is performed during a routine exam and takes between 5-10 minutes to perform. The TAEUS®-FLIP system has the potential to bring wide access to accurate liver fat measurements to a wide range of patient populations and to address the unmet need for detecting and monitoring patients with fatty liver disease and metabolic syndrome.

In this study, the investigators want to compare TAEUS® FLIP with MRI-PDFF to gain insight into the potential of thermoacoustic methods to assess liver fat content, similar to MRI-PDFF. Unlike conventional quantitative ultrasound methods, the thermoacoustic approach has demonstrated the potential to obtain estimates of liver fat fraction in individuals with high BMI (45), and those with confirmed liver fibrosis.

ELIGIBILITY:
Inclusion Criteria:

* Study participants are 18-70 years of age
* Existing MRI-PDFF not older than 6 weeks or routine MRI-PDFF in the following 6 weeks
* Be able to understand, read, and provide written informed consent in German
* Tolerant to ultrasound and MRI examinations
* Able to lay flat for 20 minutes

Exclusion Criteria:

* Metal or electronic implants, including, but not limited to: pacemakers, metal clips, drug delivery pumps, hip implants, and neural stimulation devices.
* Known pregnancy the day of consent, or becoming pregnant during study participation
* Liver disease other than NAFLD/NASH including, but not limited to, hepatitis, cirrhosis, hepatocellular carcinoma.
* Patients with broken, or injured skin, in the right upper abdominal quadrant.
* BMI over 43 kg/m2

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients referred to radiology for abdominal imaging and suspected of having steatotic liver disease.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2024-06-21 (Estimated); Primary Completion 2025-06-21 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
Thermoacoustic Fat Measurements | May 2024 to September 2025
  Perform thermoacoustic fat measurements for 80 participants, by one or more qualified operators, over the span of the study in order to determine the correlation of thermoacoustic derived fat fraction measures of steatotic liver disease to measurements obtained by MRI-PDFF.
Estimate Accuracy of Thermoacoustic Fat Fraction | May 2024 to September 2025
  Estimate the accuracy of thermoacoustic derived fat fraction measurements of steatotic liver disease by comparing to the established standard of MRI-PDFF measurements of liver fat fraction

SECONDARY OUTCOMES:
Usability Metric | May 2024 to January 2025
  To derive usability in terms of exam failure rate, where a single exam failure is defined as a failure to produce a fat fraction value for the subject. Multiple qualified users will be trained to operate, and evaluate, the TAEUS® FLIP system usability.
Estimate Operator Variability | May 2024 to January 2025
  Estimate the intra- and inter- operator variability of thermoacoustic derived liver fat fraction in 10 participants, by acquiring fat fraction measurements in replicate, by multiple operators.

CONTACTS AND LOCATIONS:
Locations (1):
- Klinikum der Universität München Großhadern Klinik und Poliklink für Radiologie, München, Germany

IPD SHARING:
Plan to Share IPD: Undecided
Data sharing is contingent on the data sharing policy of principal investigator and the study site.